CLINICAL TRIAL: NCT04015349
Title: Clinical Condition and Sleep Quality Factors Associated With Sleep Bruxism in Adults: a Study Using Polysomnography.
Brief Title: Clinical Condition and Sleep Quality Factors Associated With Sleep Bruxism in Adults.
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Associate Professor, Federal University of Pelotas
Other Study IDs: FUPelotas5
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Sleep Bruxism, Adult
Keywords: grind; polysomnography; rhythmic masticatory muscle activity; sleep bruxism
MeSH Terms: conditions — Sleep Bruxism | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography — The polysomnography (referred to as type I) allows assessing several sleep physiologic parameters (eg, EEG, electrooculogram, electromyogram, electrocardiogram, airflow, respiratory effort, oxygen saturation), whereas audio-video recording enables documenting tooth-grinding sounds and distinguishing between rhythmic masticatory muscle activity (RMMA) and orofacial (eg, swallowing) and other muscular activity (eg, head movements) during sleep. Based on the RMMA index (number of episodes per hour of sleep), sleep bruxism is diagnosed when RMMA episodes are greater than or equal to 2 (low-frequency SB, mild bruxism) or RMMA episodes are greater than or equal to 4 (high-frequency SB, severe bruxism)

SUMMARY:
This cross-sectional study will evaluate the association between sociodemographic, occupational, clinical conditions, psychological (sense of coherence), sleep quality variables and SB diagnosed by PSG, the gold standard exam with audio-visual resources obtained at Pelotas Sleep Institute.

DETAILED DESCRIPTION:
Sleep bruxism is defined as a masticatory muscle activity during sleep that is characterised as rhythmic (phasic) or non-rhythmic (tonic) and should be considered a risk factor rather than a disorder in otherwise healthy individuals.

The diagnosis of sleep bruxism often is challenging and despite the use of questionnaires, clinical exams and portable devices, based on current knowledge, the polysomnography with audio-video recordings emerges as the gold-standard criteria for a definite sleep bruxism diagnosis.

Included on the questionnaire there is a registration form, which contains: included: age at time of data collection , gender, marital status , and education level ; Occupational: individuals were asked about work outside home, and working hours; Clinical condition: body mass index, smoking; alcohol consumption; use of sleeping pills; respiratory allergy and Psychological: sense of coherence .

ELIGIBILITY:
Inclusion Criteria:

* All adults (aged 20 to 60 years) and elderly (aged >60 years)

Exclusion Criteria:

* Inadequate cognitive capacity to understand and answer the questionnaires;
* Degraded PSG image quality;
* Questionnaires filled incorrectly;
* Participants who presented a history of epilepsy that could interfere in the results of polysomnography.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All records obtained from adults (aged 20 to 60 years) and elderly (aged >60 years) who had undergone PSG at a private medical outpatients clinic from July 2017 to February 2018 were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Patients with Sleep Bruxism by Polysomnography exams | 4 months
  The data were obtained from polysomnography records in which masseter electromyography (EMG) burst was detected based on a predefined EMG threshold (20% of maximal voluntary tooth clenching task). Right masseter EMG bursts exceeding 0.25 second in duration were selected for oromotor activity scoring according to published criteria. Oromotor episodes separated by 3-second intervals were recognized as rhythmic masticatory muscle activity (RMMA) if they corresponded to 1 of the 3 following patterns: phasic (3 or more EMG bursts, each lasting 0.25 to 2 seconds), tonic (1 EMG burst lasting more than 2 seconds), or mixed (both burst types) episodes. EMG bursts were considered within the same RMMA episode if the interval between them was shorter than 2 seconds. Participants had SB diagnosed by polysomnography (PSG) if the RMMA index was greater than 2 episodes per hour of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided